CLINICAL TRIAL: NCT06568536
Title: Measuring Brain Complexity to Detect and Predict Recovery of Consciousness in the ICU (COMPASS)
Brief Title: Measuring Brain Complexity to Detect and Predict Recovery of Consciousness in the ICU
Acronym: COMPASS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Brian L. Edlow, M.D., Director, Laboratory for NeuroImaging of Coma and Consciousness (NICC), Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024P001805; 1R01NS138257-01 (NIH)
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Consciousness Disorders
Keywords: unresponsive wakefulness syndrome; vegetative state; minimally conscious state; transcranial magnetic stimulation; electroencephalography; traumatic brain injury; coma recovery scale - revised; functional electroencephalogram; functional imaging
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: The presence of consciousness will be classified considering the highest level of consciousness revealed by repeated behavioral examinations, functional electroencephalography (task-based EEG), and functional brain imagery (task-based fMRI). Based on the results of this composite standard reference, we will evaluate the diagnostic and prognostic accuracy of TMS-EEG measurements of brain complexity
Masking Description: Of note, while this is not a "multi-arm" randomized controlled trial, the outcome assessor for the 6-month functional outcome will be blinded to the patient's level of consciousness that was assessed in the ICU.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with acute disorders of consciousness receiving TMS-EEG (Experimental): Adults with acute severe traumatic brain injury who undergo advanced neuroimaging and electrophysiological studies while in the intensive care unit and are followed for 6 months post-injury.
  Interventions: Other: Repeated behavioral assessments, functional electroencephalography and brain imagery, TMS-EEG

INTERVENTIONS:
Other: Repeated behavioral assessments, functional electroencephalography and brain imagery, TMS-EEG — The presence of consciousness will be classified considering the highest level of consciousness revealed by repeated behavioral examinations, functional electroencephalography (task-based EEG), and functional brain imagery (task-based fMRI). Based on the results of this composite standard reference, we will evaluate the diagnostic and prognostic accuracy of TMS-EEG measurements of brain complexity

SUMMARY:
Disorders of consciousness (DoC) caused by severe brain injury affect millions of people worldwide each year. A patient's level of consciousness in the intensive care unit (ICU) significantly impacts the recovery from disability and is a primary determinant of family decisions about withdrawal of life-sustaining therapy (WLST). However, reliable assessment of consciousness in the ICU remains elusive. Transcranial magnetic stimulation-electroencephalography (TMS-EEG) is a tool that has shown the best performance in detecting signs of consciousness in patients with chronic DoC. The goals of this prospective, observational study are to demonstrate the diagnostic performance and prognostic utility of TMS-EEG in the ICU setting.

DETAILED DESCRIPTION:
Disorders of consciousness (DoC) caused by severe brain injury affect millions of people worldwide each year. A patient's level of consciousness in the intensive care unit (ICU) significantly influences the recovery from disability and may affect family decisions about withdrawal of life-sustaining therapy (WLST). Transcranial magnetic stimulation-electroencephalography (TMS-EEG) has shown the best performance in detecting signs of consciousness in patients with chronic DoC. The goals of this multi-center observational study are to demonstrate the diagnostic performance and prognostic utility of TMS-EEG in patients with DoC caused by severe brain injuries in the ICU.

Through this research, we aim to demonstrate that:

* TMS-EEG can detect 95% of conscious patients who are defined as conscious by a combination of tests that aim to detect overt and covert consciousness.
* TMS-EEG measurements can predict 6-month outcomes on the Disability Rating Scale (DRS) in patients in an acute vegetative state, controlling for age, Glasgow Coma Scale (GCS) score, and injury mechanism

All participants will undergo repeated behavioral assessments, task-based electroencephalography (EEG), and TMS-EEG. Of note, conventional brain magnetic resonance imaging (MRI) and task-based functional MRI are optional.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18
2. Functionally independent at baseline
3. Acquired brain injury within the last 28 days
4. Disorder of consciousness, as defined by no instance of following commands (i.e., Glasgow Coma Scale motor score = 6) on two or more consecutive assessments
5. Continuous intravenous sedation able to be discontinued for at least 10 minutes
6. ICU clinicians approve safe placement of 64-electrode EEG cap on the scalp

Additional inclusion criteria are present in the study protocol.

Exclusion Criteria:

1. Status epilepticus or uncontrolled seizure disorder
2. No head CT scan from current hospital admission AND contraindications for MRI: conductive, ferromagnetic, or other magnetic-sensitive metals implanted in the head (e.g., cochlear implants, implanted electrodes/stimulators, aneurysm clips or coils, stents, bullet fragments)
3. Medical instability, restlessness, or other factors identified by the PI that would either prevent safe participation or compromise data acquisition
4. Hemicraniectomy

If a subject meets a contraindication for MR imaging, the subject may participate in all other aspects of the study except MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Presence of consciousness as defined by a composite reference standard for consciousness that combines behavior, task-based EEG, and task-based fMRI | 48 hours after the end of the TMS-EEG assessment
  Behavioral assessments of consciousness (up to 5): The CRS-R consists of 6 subscales designed to assess auditory function, receptive and expressive language, visuoperception, communication ability, motor functions, and arousal level. The lowest score on each sub-scale represents reflexive activity; the highest represents behaviors mediated by cognitive input. The total score ranges between 0 (worst) and 23 (best). The CRSR-FAST assesses only those CRS-R behaviors that differentiate conscious (i.e., MCS) from unconscious (i.e., coma/VS) patients.
  Functional assessments of covert consciousness: A participant is classified as being conscious on task-based EEG if the probability with which the classifier distinguished task from rest conditions is p < 0.05 and the accuracy value that indicates the classifier's performance is ≥ 60%. A participant is classified as being conscious on task-based fMRI if there is one statistical activation within a pre-specified region of interest.
Disability Rating Scale (DRS) total score | 6 months post injury
  The Disability Rating Scale (DRS) provides quantitative information regarding functional disability in patients recovering from severe brain injury. The total score on the DRS ranges from 0 to 29 with higher scores indicating a greater degree of disability. DRS subscale scores include eye opening [score range 0-3], communication [score range 0-4], motor response [score range 0-5], cognitive ability for feeding [score range 0-3], cognitive ability for toileting [score range 0-3], cognitive ability for grooming [score range 0-3], level of function [score range 0-5], and employability [score range 0-3]. Subscale scores are summed to produce the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Brian L. Edlow, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - UW Health University Hospital, Madison, Wisconsin